CLINICAL TRIAL: NCT04300413
Title: Patient-Centered, Interprofessional Approach to Improve Functional Outcomes in a Skilled Nursing Facility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-2490
Record Dates: First submitted 2020-02-24; First posted 2020-03-09 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Physical Disability
MeSH Terms: interventions — Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: This is a single arm study but will use two historical cohorts as comparison groups to assess outcomes: 1) usual care and 2) high-intensity, functionally based resistance training alone. The historical cohorts were included in a previous study (Clinical Trials Registry identifier: E2193-P). This design will include independent cohorts of patients within a single SNF, using the facility as its own control. This design optimally controls for facility-level variables that vary widely between SNFs and may influence care delivery, such as staffing levels, staff experience, and productivity standards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Intensity Rehabilitation plus Mobility (HeRo) (Experimental): The HeRo group will receive a behavior-change intervention based in the principals of behavioral economics to improve mobility. Physical and occupational therapists have been trained to deliver a high-intensity, functional intervention as the standard of care in this skilled nursing facility.
  Interventions: Other: High-Intensity Rehabilitation plus Mobility (HeRo)

INTERVENTIONS:
Other: High-Intensity Rehabilitation plus Mobility (HeRo) — Progressive, high-intensity strengthening and functional intervention coupled with structured mobility based in principals of behavioral economics.

SUMMARY:
During a hospital stay, older adults often become physically deconditioned and lose their ability to perform activities of daily living. Afterwards, they commonly require rehabilitation in a skilled nursing facility to regain independence. Even at discharge, however, many older adults are still far below their pre-hospitalization level of function making them at risk for adverse events such as falls, rehospitalizations, and loss of independence. Two reasons for inadequate outcomes may include that 1) physical and occupational therapy interventions are delivered at too low an intensity to incur substantial physiological gains, and 2) residents are largely sedentary outside of structured therapy time. These two problems represent critical targets for interventions that optimize care in skilled nursing facilities. Therefore, the investigators designed High-Intensity Rehabilitation + Mobility (HeRo), a patient-centered approach to skilled nursing facility care that incorporates a combination of high-intensity (i.e. high resistance, low repetition) functionally-based resistance training along with a structured mobility program outside of therapy time.

HeRo includes: 1) a team approach to patient-centered care; 2) a physical activity intervention that incorporates principals of behavioral economics, which uses incentives, goal setting, and gamification to optimize patient engagement and health outcomes and 3) a challenging, high-intensity rehabilitation intervention that pushes patients to expand their limits. The investigators expect that HeRo will improve physical function and physical activity while reducing sedentary time for older adults in the skilled nursing facility. The study team will assess the feasibility and acceptability of HeRo for multiple stakeholders including patients, physical and occupational therapists, nursing staff, and administration. This research will improve patient care in the skilled nursing facility environment, getting older adults on a fast track to developing independence after a hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 50 who are admitted to a skilled nursing facility following hospitalization
* Qualify to receive at least physical therapy services
* Ambulatory prior to hospitalization

Exclusion Criteria:

1. Patients with neurological disorders such as acute stroke or acute traumatic brain injury
2. Patients on hospice care
3. Patient with conditions where strength training is contraindicated (as indicated by the American College of Sports Medicine Guidelines for Exercise Testing and Prescription):

   1. Recent unstable fracture
   2. Advanced congestive heart failure
   3. Bone metastasis sites
   4. Tumors in strengthening target areas
   5. Acute Illness
   6. Recent myocardial infarction (within 3-6 weeks)
   7. Weight bearing restrictions on graft or fracture sites
   8. Exposed tendon or muscle
   9. Absence of pedal pulses
   10. Presence of fistula
   11. Platelet levels <50,000/μL
4. Weight-bearing precautions and inability to ambulate prior to hospitalization

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-02-16 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Gait Speed | Change from date of admission into the SNF to date of discharge from the SNF, which would be an approximate average of 21 days
  Time it takes to walk 4 meters (meters per second)

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Change from date of admission into the SNF to date of discharge from the SNF, which would be an approximate average of 21 days
  Global measure of lower extremity function, which consists of walking speed, chair stands, and balance tests

OTHER OUTCOMES:
Patient Satisfaction Survey | At date of discharge after their stay in the Skilled Nursing Facility, (approximately 21 days after admission).
  8 question survey on patient satisfaction, scoring each question on a 1-10 scale (1=not at all and 10=extremely)
Physical Activity (upright time) | Measured during the last 5 days before discharge date from Skilled Nursing Facility (approximate average length of stay 21 days).
  Percent waking hours spent upright measured using ActivPAL devices
Physical Activity (sedentary time) | Measured during the last 5 days before discharge date from Skilled Nursing Facility (approximate average length of stay 21 days).
  Time spent in sedentary bouts measured using ActivPAL devices
Treatment fidelity | At least 2 observations per provider per year throughout duration of study (approximately 2 years), 2 additional observations scheduled if compliance is <80% on objective fidelity checklist.
  Provider intervention compliance with high-intensity rehabilitation (PT and OT) and mobility (nursing staff) using a fidelity checklist

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevens-Lapsley, PT, PhD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Veterans Community Living Center at Fitzsimmons, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mallinson T, Deutsch A, Bateman J, Tseng HY, Manheim L, Almagor O, Heinemann AW. Comparison of discharge functional status after rehabilitation in skilled nursing, home health, and medical rehabilitation settings for patients after hip fracture repair. Arch Phys Med Rehabil. 2014 Feb;95(2):209-17. doi: 10.1016/j.apmr.2013.05.031. Epub 2013 Jul 10. PMID 23850612
- [Background] Simning A, Caprio TV, Seplaki CL, Temkin-Greener H, Szanton SL, Conwell Y. Patient-Reported Outcomes in Functioning Following Nursing Home or Inpatient Rehabilitation. J Am Med Dir Assoc. 2018 Oct;19(10):864-870. doi: 10.1016/j.jamda.2018.06.014. Epub 2018 Jul 25. PMID 30056009
- [Background] Grant PM, Granat MH, Thow MK, Maclaren WM. Analyzing free-living physical activity of older adults in different environments using body-worn activity monitors. J Aging Phys Act. 2010 Apr;18(2):171-84. doi: 10.1123/japa.18.2.171. PMID 20440029

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT04300413/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT04300413/ICF_001.pdf